CLINICAL TRIAL: NCT04289870
Title: Prospective, Single Arm, Multi-center, First-in-human (FIH) Study to Assess the Safety and Performance of the Innoventric Trillium™ Stent Graft for the Treatment of Severe Tricuspid Regurgitation (TR)
Brief Title: Innoventric Trillium™ Stent Graft First-in-Human (FIH) Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Innoventric LTD (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLD-001
Record Dates: First submitted 2020-02-05; First posted 2020-02-28 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Tricuspid Regurgitation
Keywords: Tricuspid Valve; Tricuspid Valve Insufficiency; Tricuspid Regurgitation
MeSH Terms: conditions — Tricuspid Valve Insufficiency

STUDY DESIGN:
Intervention Model Description: First In Human study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Innoventric Trillium™ Stent Graft Single Arm (Experimental): Single-arm, open label, multi-center study
  Interventions: Device: Trillium™

INTERVENTIONS:
Device: Trillium™ — Trillium™ Stent Graft for Functional Tricuspid Valve Replacement

SUMMARY:
A prospective, single-arm, multi-center first-in-human (FIH) study to evaluate the safety and performance of the Innoventric Trillium™ Stent Graft System.

Twenty (20) patients in 8 investigational sites will be enrolled. All enrolled study patients will be assessed at baseline, during the procedure, at discharge, after 1 month, 3 months, 6 months, 1 year, 1.5 years, 2 years, and 3 years following the index procedure.

ELIGIBILITY:
Inclusion Criteria:

Enrolled patients must meet ALL the following criteria:

1. Age >40 (no upper limit)
2. Patient has clinically significant TR graded as severe based on the presence of systolic hepatic vein flow reversal, and VCW≥7mm or EROA≥40mm^2
3. Symptomatic despite medical therapy; patient must be on diuretic therapy.
4. Peak central venous pressure of ≥ 15mmHg
5. The local site Heart Team determines that the patient is appropriate for transcatheter tricuspid intervention
6. Patient is willing and able to comply with all specified study evaluations.
7. Patient has NYHA functional classification of III or IV
8. Patient is not eligible for standard-of-care surgical or interventional therapy assessed by the central heart team or has refused standard-of-care surgical and interventional therapy or has received standard-of-care TR therapy and remains symptomatic
9. Patient understands the nature of the study and study requirements and is willing to provide written Informed Consent prior to any study-specific procedures.

Exclusion Criteria:

Patients will be excluded from participation if ANY of the following criteria apply:

1. Echocardiographic parameters (Any of the following):

   I. LVEF < 20% II. Evidence of severe right ventricular dysfunction (e.g. right ventricular TAPSE < 13.0mm) III. IVC or SVC anatomy that precludes proper device deployment and function
2. Systolic Pulmonary Artery Pressure > 70mmHg
3. Severe aortic, mitral, and/or pulmonic valve stenosis and/or regurgitation
4. Active endocarditis within 90 days of the scheduled implant
5. Significant pericardial effusion
6. Intra-cardiac masses, thrombi, or vegetation
7. Thrombosis of the venous system
8. Space-consuming lesion in the heart or on the valves, thrombus, or microbial colonization of the valves
9. Untreated clinically significant coronary artery disease requiring immediate revascularization
10. MI or known unstable angina within 30 days prior to the index procedure
11. Any therapeutic invasive cardiac procedure within 30 days prior to the index procedure
12. Any prior cardiac surgery, within 3 months of the index procedure
13. Hemodynamic instability or treated with IV inotropes within 30 days of the index procedure
14. Severe uncontrolled hypertension (SBP ≥ 180 mmHg and/or DBP ≥ 110 mm Hg)
15. Severe uncontrolled hypotension (SBP≤80 mmHg and/or DBP≤40 mmHg)
16. Cerebrovascular Accident (CVA) within the past 90 days
17. Kidney dysfunction with estimated Glomerular Filtration Rate (eGFR) < 30 ml/min/1.73 m^2 or patient is on chronic dialysis
18. Significant frailty (i.e. Clinical Frailty Scale© (CFS) ≥ 7) within 90 days of the scheduled implant procedure
19. Chronic liver disease with a MELD score of 20 or greater
20. Chronic anemia (Hb < 9 g/L) not corrected by transfusion
21. Thrombocytopenia (Platelet count< 100,000/mm3) or thrombocytosis (Platelet count > 750,000/mm3)
22. Bleeding disorders or hypercoagulable state
23. Active peptic ulcer or active gastrointestinal (GI) bleeding within 90 days of the scheduled implant
24. Contraindication to anticoagulants or antiplatelet agents
25. Currently or history of IV drug use
26. Pregnant or lactating; or female of childbearing potential with a positive pregnancy test 24 hours before any study-related radiation exposure.
27. Inability to access the femoral vein with a 24 FR guide (e.g., DVT, occluded femoral veins).
28. Known allergy to stainless steel, nickel, titanium, PET or contrast agents that cannot be adequately pre-medicated.
29. Known hypersensitivity or contraindication to procedural medications which cannot be adequately managed medically
30. Impaired judgment
31. Undergoing emergent or urgent treatment for tricuspid insufficiency
32. Currently participating in another investigational drug or device study that has not completed the primary endpoint or that clinically interferes with the endpoints of this study
33. Co-morbid condition(s) that, in the opinion of the Investigator, limit life expectancy to < 12 months
34. Cardiac cachexia
35. In the judgment of the Investigator, co-morbid condition(s) that could limit the patient's ability to participate in the study, including compliance with follow-up requirements, or that could impact the scientific integrity of the study
36. Patient is under guardianship
37. Presence of any prosthetic device in the SVC or IVC (excluding pace-maker, ICD and CRT leads)
38. Elevated inflammatory markers within 2 weeks of the scheduled procedure (e.g. CRP>1.5mg/dL).

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-06-24 (Actual); Primary Completion 2023-07-21 (Actual); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Safety Endpoint | Evaluated immediately after intervention, discharge and 30 days
  Rate of device or procedure-related MAEs
  and
  Freedom from unplanned surgery or re-intervention, due to life-threatening device or procedure failure
Technical performance | Evaluated immediately after intervention
  Successful access, delivery, and retrieval of the Trillium delivery system, the device is anchored both in SVC and IVC.
Efficacy Endpoint | Evaluated immediately after intervention
  TR grade as measured on the device valves (Echocardiography), or by hepatic vein systolic backflow (Echocardiography), or reduction in peak central venous pressure (Invasive hemodynamic measurement).

SECONDARY OUTCOMES:
Safety Endpoint | Assessment at 3-month, 6-month and 1-year
  Composite of all device or procedure-related MAEs.
Efficacy Endpoint | Assessment at 30 days, 3-month, 6-month and 1-year
  One or more of the following-
  * TR grade measured on the device valves (Echocardiography), or by hepatic vein systolic backflow (Echocardiography), or measured by a regurgitant fraction (CMR) [at 30 days, 3-month, 6-month, and 1-year]
  * Rate of hospitalizations for HF [at 30 days, 3-month, 6-month, and 1-year]
  Or one or more of the following-
  * Clinical Frailty Scale (CFS) [at 30 days, 3-month, 6-month, and 1-year]
  * HF functional class (NYHA) [at 30 days, 3-month, 6-month, and 1-year]
  * Six-minute walk test (6MWT) [at 30 days, 3-month, 6-month, and 1-year]
  * The Kansas City Cardiomyopathy Questionnaire (KCCQ) [at 30 days, 3-month, 6-month, and 1-year]

OTHER OUTCOMES:
Other Endpoints | Assessment at 30 days, 3-month, 6-month and 1-year
  transthoracic echocardiography (TTE) will be performed to determine acceptable performance of the device defined as a reduction in hepatic vein systolic backflow to moderate (systolic blunting) or better. In addition, the tricuspid valve complex will be imaged to capture the following parameters for comparison to baseline: Page 46 of 118 -Confidential-
  1. TR grade (qualitative)
  2. Jet area
  3. EROA and regurgitant volume
  4. RV and LV dimensions
  5. RA area/volume
  6. LVEF
  7. Tricuspid annular plane systolic excursion (TAPSE)
  8. IVC dimensions/respiratory variations
  9. Pulmonary artery pressure (PAP)
  10. Right atrial pressure (RAP)
  11. RV pressure
  12. IVC/SVC pressure It should be noted that the above-mentioned parameters are primarily being captured for research purposes and may not be affected by the device.
  The following clinical and laboratory parameters will be captured for comparison to baseline values:
  1. Mini Nutrition Assessment (MNA)®
  2. Clinical Frailty Scale©

CONTACTS AND LOCATIONS:
Locations (9):
- Belgium (2):
  - OLVZ Aalst, Aalst
  - ZNA, Antwerp
- Germany (3):
  - Heart & Diabetes Center NRW, Bad Oeynhausen
  - Herzzentrum der Charité (DHZC), Berlin
  - Leipzig Heart Center, Leipzig
- Rabin Medical Center, Petah Tikva, Israel
- Spain (3):
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Universitario de Salamanca, Salamanca
  - Hospital Alvaro Cunqueiro, Hospital Universitario de Vigo, Vigo

IPD SHARING:
Plan to Share IPD: Undecided